CLINICAL TRIAL: NCT05557123
Title: The ReInforcement of Adherence Via Self-monitoring App Orchestrating Biosignals and Medication of RivoXaban in Patients with Atrial Fibrillation and Co-morbidities: Randomised Control Study(RIVOX-AF Study)
Brief Title: Mobile App for Improving Adherence of Rivoxaban (RIVOX-AF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: SAMJIN PHARM (Unknown)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIVOX-AF
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; mobile app
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEDI-app (Experimental): conventional treatment with MEDI-app feedback
  Interventions: Device: MEDI-app
- conventional treatment (No Intervention): conventional treatment

INTERVENTIONS:
Device: MEDI-app — MEDI-app based feedback algorithm. The app based feedback algorithm will check and remind the patients of taking medication.
  Arms: MEDI-app

SUMMARY:
RIVOX-AF study is a prospective, multicenter, randomized controlled study in which patients with AF are allocated to medication-app group or conventional treatment group. The App based feed-back algorithm will provide the patients with check taking drug or reminding of taking drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AF aged 19 years or older with one or more comorbidities including heart failure, myocardial infarction, stable angina, hypertension or diabetes mellitus (Patients can be enrolled 3 months after myocardial infarction or percutaneous coronary intervention).
* patients who already took or plan to take rivoxban
* patients who able to use smart phone

Exclusion Criteria:

* creatinine clearance <15ml/min
* moderate or severe mitral stenosis
* mitral valve operation history
* current alcohol abuse or alcohol abus history
* Not eligible for study due to legal or psychiatric problem
* enrolled other clinical study within 4 weeks
* declined to enroll the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Drug adherence | 24 week
  Drug adherence by pill count
Proportion of adequate medication adherence at 24 weeks | 24 weeks
  proportion of patients with ≥95% of continuous medication adherence

SECONDARY OUTCOMES:
The occurrence of clinical composite end point | 24 week
  composites of stroke, systemic embolic event, major bleeding requiring hospitalization or transfusion, or death.)
The occurrence of MACCE and hospitalization | 24 week
  MACCE plus hospitalization
The occurrence of Thromboembolism (Stroke, TIA, Pulmonary embolism) | 24 week
  Stroke, TIA, Pulmonary embolism)
The occurrence of bleeding | 24 week
  bleeding event
Drug adherence | 12 week
  Drug adherence by pill count
Proportion of adequate medication adherence at 12 weeks | 12 week
  proportion of patients with ≥95% of continuous medication adherence
medication adherence by zero-inflated model | 12 week and 24 weeks
  medication adherence by zero-inflated model

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD, PhD, Study Chair — Seoul National Univeristy Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Yoon M, Park JJ, Hur T, Hua CH, Shim CY, Yoo BS, Cho HJ, Lee S, Kim HM, Kim JH, Lee S, Choi DJ. The ReInforcement of adherence via self-monitoring app orchestrating biosignals and medication of RivaroXaban in patients with atrial fibrillation and co-morbidities: a study protocol for a randomized controlled trial (RIVOX-AF). Front Cardiovasc Med. 2023 May 24;10:1130216. doi: 10.3389/fcvm.2023.1130216. eCollection 2023. PMID 37324622